CLINICAL TRIAL: NCT04465097
Title: Neoadjuvant Tucidinostat and Exemestane in Estrogen Receptor-Positive Early Breast Cancer （NeoTEE）
Brief Title: Neoadjuvant Tucidinostat and Exemestane in Early Breast Cancer
Acronym: NeoTEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Lin, Vice Director of Department of Breast Surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200628GD
Record Dates: First submitted 2020-06-30; First posted 2020-07-09 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Tucidinostat; Estrogen Receptor-Positive; Neoadjuvant endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat and Exemestane (Experimental): Patients receive exemestane from week 1 to week 26 and Tucidinostat BIW from week 3 to week 26. Courses continue in the absence of disease progression or unacceptable toxicity. If the patient is premenopausal, leuprorelin or goserelin will be prescribed.
  Interventions: Drug: Tucidinostat; Drug: Exemestane; Drug: Ovarian function suppression

INTERVENTIONS:
Drug: Tucidinostat — Tucidinostat: 30 mg BIW (Monday and Thursday) from week 3 to week 26
  Other Names: Chidamide; Epidaza
Drug: Exemestane — Exemestane: 25 mg QD from week 1 to week 26.
Drug: Ovarian function suppression — If the patient is premenopausal, leuprorelin 3.75mg or goserelin 3.6 mg will be injected every 28 days.

SUMMARY:
This study is to evaluate the efficacy of tucidinostat combined with exemestane as neoadjuvant strategy in estrogen receptor-positive early breast cancer patients and explore the genetic model which can predict neoadjuvant endocrine therapeutic results.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy of tucidinostat combined with exemestane as neoadjuvant strategy in estrogen receptor-positive early breast cancer patients.This study will recruit 30 patients. The 30 patients will receive 25 mg exemestane QD for 26 weeks. Tucidinostat will be prescribed 30 mg BIW from week 3 to week 26. During neoadjuvant treatment biopsy, CEUS and MRI will be perfomed according to protocol to evaluate the therapeutic results. Genetic testing will also be performed before and after neoadjuvant treatment to explore the predictive value. MRI evaluated ORR is primary end point. CEUS evaluated ORR, pCR, AE and RCB are secondary end point.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed；
2. Eastern Cooperative Oncology Group Performance Status: 0~1;
3. Histological confirmation of estrogen receptor (ER) positive and HER 2 negative invasive breast cancer;
4. Age ≥18 years old；
5. No distant metastatic disease；
6. The disease condition is stage II or stage III;
7. Laboratory exam criteria for enrollment: HGB≥10g/dl, WBC≥4,000/mm3, PLT≥100,000/mm3, GOT, GPT, ALP≤2 times ULN, TBIL, CCr≤1.5 times ULN.

Exclusion Criteria:

1. Patients who are pregnant or lactating at the time of randomization or refuse to contraception.
2. Patients who received organ transplantation (include bone marrow autologous transplantation and stem cell transplantation).
3. Patients who have other malignant diseases within 5 years, except for cured skin basal cell carcinoma, flat cell carcinoma or cervical carcinoma in situ
4. Patients with psychiatric disorder, peripheral or central nerve system disease or any disorder, which compromises ability to give informed consent or participate in this study.
5. Patients with sever hepatic, renal,cardiovascular, respiratory, digestive diseases or uncontrolled diabetes.
6. Patients who had myocardial infarction in the past 12 months.
7. Patients who participate in other clinical trail.
8. Patients who allergy to goserelin, leuprorelin, tucidinostat or aromatase inhibitor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) evaluated by MRI | Up to 31 weeks
  ORR is defined as percentage of participants with Complete Response and Partial Response, assessed by the investigators using MRI according to the Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
objective response rate (ORR) evaluated by CEUS | Up to 31 weeks
  Contrast-enhanced ultrasound will also be performed to assess ORR
pathologic complete response rate (pCR) | Up to 31 weeks
  The percentage of participants with pathologically assessed ypT0 and ypTis of breast disease.
Adverse effect (AE) | Up to 31 weeks
  All advese effect events related with Tucidinostat and Exemestane.
Residual Cancer Burden (RCB) | Up to 31 weeks
  Pathologilly assessed residual cancer burden according to MD Anderson protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lin, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The first affiliated hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang Z, Li W, Hu X, Zhang Q, Sun T, Cui S, Wang S, Ouyang Q, Yin Y, Geng C, Tong Z, Cheng Y, Pan Y, Sun Y, Wang H, Ouyang T, Gu K, Feng J, Wang X, Wang S, Liu T, Gao J, Cristofanilli M, Ning Z, Lu X. Tucidinostat plus exemestane for postmenopausal patients with advanced, hormone receptor-positive breast cancer (ACE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Jun;20(6):806-815. doi: 10.1016/S1470-2045(19)30164-0. Epub 2019 Apr 27. PMID 31036468